CLINICAL TRIAL: NCT02586129
Title: Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Trial to Evaluate the Safety and Efficacy of YH14755 in Subjects With Dyslipidemia and Type II Diabetes
Brief Title: Clinical Trial of YH14755 in Subjects With Dyslipidemia and Type II Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH14755-301
Record Dates: First submitted 2015-09-22; First posted 2015-10-26 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Dyslipidemia; Type II Diabetes
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2 | interventions — Metformin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- YH14755 (Experimental): PO, Once Daily, 16 weeks
  Interventions: Drug: YH14755
- Metformin (Active Comparator): PO, Once Daily, 16 weeks
  Interventions: Drug: Metformin
- Rosuvastatin (Active Comparator): PO, Once Daily, 16 weeks
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: YH14755 — 20/1500mg, QD
  Arms: YH14755
Drug: Metformin — 1500mg, QD
  Arms: Metformin
Drug: Rosuvastatin — 20mg, QD
  Arms: Rosuvastatin

SUMMARY:
Randomized, double-blind, active-controlled, multicenter phase 3 trial to evaluate the safety and efficacy of YH14755 in subjects with dyslipidemia and Type II Diabetes.

DETAILED DESCRIPTION:
This is a phase 3 trial to evaluate the safety and efficacy of YH14755 in subjects with dyslipidemia and Type II Diabetes.

In YH14755 treatment group, 88 subjects will be assigned and the subjects administer YH14755 for 16 weeks.

In Metformin treatment group, 88 subjects will be assigned and the subjects administer Metformin for 16 weeks.

In Rosuvastatin treatment group, 88 subjects will be assigned and the subjects administer Rosuvastatin for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Subjects with Dyslipidemia and Type II Diabetes
* 6.5% ≤ HbA1c level ≤ 9.0% and LDL-C level ≤ 250mg/dL(6.5 nmal/L) at screening
* BMI ≤ 45kg/m2
* Subjects who dose not administered diabetes treatment at least 4 weeks prior to screening visit.
* 19 years later, men and women under the age of 75

Exclusion Criteria:

* Pregnant women, nursing mothers or subject who does not agree to assigned contraception in the study
* Subject with type I Diabetes
* Subject with hypertension which does not controlled by treatment(have blood pressure > 160/110mmHg)
* Have a known allergy to drugs
* Have administered Cyclosporine
* Have administered Obesity treatment within 12 weeks prior to screening visit
* Participated in any other clinical trials within 30 days prior to the first administration
* Subject who is judged to be ineligible by investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Change in LDL Cholesterol | Change from baseline at 16 weeks
Change in HbA1c | Change from baseline at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hakcheol Jang, M.D., Ph.D., Study Chair — Department of Internal Medicine, SNU Bundang Hospital
Locations (1):
- Seoul National Universitiy Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea